CLINICAL TRIAL: NCT06249178
Title: Developing Extracellular Vesicle Based MPRINT Translational Resource Platform for Monitoring Therapeutics Response During Pregnancy
Brief Title: EV Based Platform for Monitoring Therapeutics Response During Pregnancy (ARISE)
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: University of Texas (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maged Costantine, MD, MBA, Professor, Ohio State University
Other Study IDs: 2024H0050; 1R24HD113024 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia
Keywords: Extracellular vesicles proteome profile; Aspirin treatment; Pregnancy; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and optional placenta samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective observational cohort study of pregnant people at-risk of preeclampsia receiving aspirin as part of clinical care or a planned randomized controlled trial of 81mg vs. 162mg of aspirin is to generate proteomic data to show a distinct maternal and fetal Extracellular Vesicle (EV) proteome profile with aspirin treatment, and develop and validate a multi-marker panel for the monitoring of placental function in people at-risk of Preeclampsia and in response to aspirin treatment. The primary research question is:

1. Does the maternal and fetal Positive for Placental Alkaline Phosphatase (PLAP+) Extracellular Vesicle (EV) proteome profile in the 2nd and 3rd trimester of pregnancy differ between people who receive aspirin and develop (or not) preeclampsia?

Participants will be asked to give blood samples up to four times during and at the end of their pregnancy.

DETAILED DESCRIPTION:
Pregnant and lactating people remain therapeutic orphans as they are excluded from the vast majority of clinical drug development and therapeutic trials. Moreover, current practices in drug evaluation in pregnancy have been hindered by the lack of effective biomarkers and innovative study designs. There is a need to develop novel placental-specific biomarkers in order to assess placental function and response to therapeutics, as a way to inform on their safety and efficacy. An example of these novel biomarkers is placental (fetal) specific extracellular vesicles (EVs). Recent advances in characterizing the cargo content of these EVs demonstrated their potential to be used as placental biomarkers. Fourteen proteins found in EVs significantly correlated with aspirin use (FDR<0.1) in at-risk people, but that more power is needed to confidently assess the relationship with aspirin dosage and pregnancy outcomes. In addition, prior studies showed that aspirin affects endothelial and trophoblast cells, thus potentially modulating exosome derived from these cells and their cargo contents.

The main goal is to develop a novel platform using exosome profiling, as novel biomarkers, to monitor placental mediated adverse pregnancy outcomes and response to therapeutics.

Specific Aim 1: Develop and validate a multi-marker panel/Extracellular Vesicle (EV) proteome profile (maternal and fetal) for monitoring of placental/fetal membrane function in people at-risk of Preeclampsia (PE) and in response to aspirin treatment.

Specific Aim 2: Demonstrate that maternal and fetal Positive for Placental Alkaline Phosphatase (PLAP+) EV proteome profile in the 2nd and 3rd trimester of pregnancy differ between people who develop (or not) preeclampsia and correlate with aspirin dose and salicylic acid concentrations.

Specific Aim 3: Demonstrate that the changes in maternal and fetal EV proteome profiles (baseline to 2nd-3rd trimester) correlate with the changes in inflammatory and angiogenic imbalance profiles associated with PE, and with other clinical outcomes such as Preterm Birth (PTB) and Fetal Growth Restriction (FGR).

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible to participate if they meet the following study inclusion criteria:

1. pregnant individuals age ≥18 years
2. enrolled ≤16 6/7 weeks of gestation based on the best obstetric estimate as defined by ACOG criteria
3. singleton live intrauterine gestation
4. Any of the following:

   1. At least one of the high-risk criteria for HDP (per US Preventive Services Task Force Recommendation Statement [USPSTF]); i) any prior pregnancy complicated by Preeclampsia ii) current pregnancy complicated by chronic hypertension iii) chronic kidney disease iv) autoimmune disease (e.g., antiphospholipid syndrome, lupus) or
   2. Two or more moderate-risk criteria for HDP (per USPSTF); i) nulliparity (no prior delivery at or after 20 weeks 0 days of gestation) ii) obesity (body mass index ≥30 kg/m2 at time of enrollment) iii) age ≥35 years (at time of expected estimated due date) iv) Black race v) Low income vi) Personal risk factors (previous pregnancy with low birth weight or SGA infant, previous adverse pregnancy outcome [unexplained stillbirth], placental abruption, interval >10 years between pregnancies).

      vii) Pregnancy after in vitro conception viii) family history of preeclampsia ( i.e., mother or sister)
   3. or participating in another clinical RCT of 81mg vs. 162mg aspirin for prevention of hypertensive disorders of pregnancy

Exclusion Criteria:

1. age < 18 years,
2. involuntarily confined or detained
3. considered as having a diminished decision-making capacity
4. multifetal gestation
5. pregestational diabetes mellitus or gestational diabetes diagnosed < 20 weeks due to the impact on exosome response
6. known or suspected fetal aneuploidy or major congenital abnormality, fetal demise, or planned pregnancy termination
7. known allergy or hypersensitivity to aspirin or any medical condition where aspirin is contraindicated (e.g., peptic ulcer disease, nasal polyps, NSAID-induced asthma, gastrointestinal bleeding, G6PD deficiency, severe hepatic dysfunction, bleeding disorders)
8. plan to deliver at another center or participating in another intervention study that influences the primary outcome in this study, without prior approval

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women greater than 18 years of age at risk of preeclampsia (PE), receiving aspirin to prevent PE or a candidate to receive aspirin.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
multi-marker panel | From enrollment till delivery; up to 29 weeks
  Multi-marker panel (list of proteins) associated with placental function in people at-risk of PE and in response to aspirin treatment.

SECONDARY OUTCOMES:
Preeclampsia | From enrollment to deliver; up to 29 weeks
  Preeclampsia defined according to ACOG guidelines
Preterm birth < 37 weeks gestation | From enrollment to deliver; up to 25 weeks
  Delivery before 37 0/7 weeks gestation
Preterm birth < 34 weeks gestation | From enrollment to deliver; up to 22 weeks
  Delivery before 34 0/7 weeks gestation
Preeclampsia with severe features | From enrollment to deliver; up to 29 weeks
  Preeclampsia with severe features as defined by the ACOG diagnostic criteria
Gestational hypertension | From enrollment to deliver, up to 29 weeks
  Gestational hypertension defined as new onset hypertension in the absence of accompanying proteinuria or other features of preeclampsia
Fetal growth restriction | From enrollment to deliver; up to 29 weeks
  Estimated fetal weight or abdominal circumference <10%
Birthweight | at delivery
  weight of newborn at time of birth
PlGF | 28 to 41 weeks
  Serum concentration of PlGF in the third trimester
sFLT-1 | 28 to 41 weeks
  Serum concentration of sFLT-1 in the third trimester

CONTACTS AND LOCATIONS:
Overall Officials: Maged Costantine, MD, MBA, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No